CLINICAL TRIAL: NCT01086033
Title: A 3-year Post-marketing Observational Study Following up Patients With Moderate to Severe RA Treated With Humira in Greece
Brief Title: A 3-year Study Following up Patients With Moderate to Severe Rheumatoid Arthritis Treated With Humira in Greece
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: PMOS GREC 2004 06
Record Dates: First submitted 2010-02-26; First posted 2010-03-12 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Evaluation of safety and efficacy; Adalimumab treatment; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Humira: Participants with rheumatoid arthritis treated with Humira (adalimumab) as prescribed by the rheumatologist in the setting of routine clinical care.

SUMMARY:
The objectives of the study are to observe and assess the long-term use, safety and efficacy of Humira (adalimumab), as prescribed by the rheumatologist in a normal clinical setting and in accordance with the terms of the European marketing authorization and to observe compliance of patients with the prescribed treatment.

DETAILED DESCRIPTION:
This is a multi-center, uncontrolled observational study of patients who at the time of entry had moderate to severe rheumatoid arthritis (RΑ) and who were subsequently prescribed Humira (adalimumab) following normal clinical practice, with or without other anti-rheumatic treatments, prior to enrollment in this study.

Once the physician has determined that the patient meets the inclusion criteria, and the patient has agreed to be included in the observational study by signing the informed consent, the patient's Day 1 demographic data, and disease status will be reported in the Day 1 Data Report Forms. The physician will then follow-up with the patient via regular office visits at intervals as determined by routine clinical practice. Patient's safety and efficacy data, if they are part of clinical routine, will be recorded in the Data Report Forms at Day 1, and regular visits which are closest to Month 3, Month 6, Month 9, Month 12, Month 18, Month 24, Month 30, and Month 36.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate or severe active rheumatoid arthritis, who have been prescribed and are receiving Humira (adalimumab) under normal clinical practice for at least one month prior to inclusion and according to the approved Summary of Product Characteristics (SPC) in the European Union.
* Patients must be willing to consent to data being collected and provided to Abbott Laboratories.

Exclusion Criteria:

* Contraindications according to the SPC.
* Patients should not participate in another observational Abbott study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis on Humira (adalimimab) treatment
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2006-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanasis Floros, MD, Study Chair — AbbVie Pharmaceuticals S.A.
Locations (60):
- Greece (60):
  - Site Reference ID/Investigator# 30116, A. Glyfada
  - Site Reference ID/Investigator# 47544, Ag. Dimitrios, Athens
  - Site Reference ID/Investigator# 47542, Ag. Paraskevi, Athens
  - Site Reference ID/Investigator# 29915, Alexandroupoli
  - Site Reference ID/Investigator# 30118, Arta
  - Site Reference ID/Investigator# 29989, Athens
  - Site Reference ID/Investigator# 29914, Athens
  - Site Reference ID/Investigator# 29950, Athens
  - Site Reference ID/Investigator# 5284, Athens
  - Site Reference ID/Investigator# 29944, Athens
  - Site Reference ID/Investigator# 30474, Athens
  - Site Reference ID/Investigator# 29953, Athens
  - Site Reference ID/Investigator# 30085, Athens
  - Site Reference ID/Investigator# 30472, Athens
  - Site Reference ID/Investigator# 30479, Athens
  - Site Reference ID/Investigator# 30480, Athens
  - Site Reference ID/Investigator# 29899, Athens
  - Site Reference ID/Investigator# 30178, Athens
  - Site Reference ID/Investigator# 30785, Athens
  - Site Reference ID/Investigator# 30788, Athens
  - Site Reference ID/Investigator# 29992, Ágioi Anárgyroi
  - Site Reference ID/Investigator# 29954, Ágioi Anárgyroi
  - Site Reference ID/Investigator# 30198, Chalcis
  - Site Reference ID/Investigator# 30789, Cholargós
  - Site Reference ID/Investigator# 30008, Crete
  - Site Reference ID/Investigator# 30210, Crete
  - Site Reference ID/Investigator# 29828, Crete
  - Site Reference ID/Investigator# 30105, Drama
  - Site Reference ID/Investigator# 29820, Elefsina
  - Site Reference ID/Investigator# 30146, Ermoupolis Syros
  - Site Reference ID/Investigator# 30767, Heraklion Crete
  - Site Reference ID/Investigator# 30482, Ioannina
  - Site Reference ID/Investigator# 47322, Karditsa
  - Site Reference ID/Investigator# 29850, Katerini
  - Site Reference ID/Investigator# 30189, Kavala
  - Site Reference ID/Investigator# 30476, Kifissia
  - Site Reference ID/Investigator# 30004, Kozani
  - Site Reference ID/Investigator# 29993, Lamia
  - Site Reference ID/Investigator# 30770, Larissa
  - Site Reference ID/Investigator# 29988, Larissa
  - Site Reference ID/Investigator# 29922, Nikaia
  - Site Reference ID/Investigator# 29972, Pátrai
  - Site Reference ID/Investigator# 29916, Pátrai
  - Site Reference ID/Investigator# 29827, Peristeri
  - Site Reference ID/Investigator# 29936, Pýrgos
  - Site Reference ID/Investigator# 30200, Rion, Patras
  - Site Reference ID/Investigator# 29900, Thessaloniki
  - Site Reference ID/Investigator# 30192, Thessaloniki
  - Site Reference ID/Investigator# 30165, Thessaloniki
  - Site Reference ID/Investigator# 30765, Thessaloniki
  - Site Reference ID/Investigator# 29845, Thessaloniki
  - Site Reference ID/Investigator# 30791, Thessaloniki
  - Site Reference ID/Investigator# 30792, Thessaloniki
  - Site Reference ID/Investigator# 47543, Thessaloniki
  - Site Reference ID/Investigator# 29924, Thessaloniki
  - Site Reference ID/Investigator# 30477, Thessaloniki
  - Site Reference ID/Investigator# 29947, Thessaloniki
  - Site Reference ID/Investigator# 30115, Trikala
  - Site Reference ID/Investigator# 30084, Véria
  - Site Reference ID/Investigator# 29968, Xánthi

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Humira
Started | 566
Completed | 262
Not Completed | 304
Not completed — Lack of efficacy/Exacerbation of RA | 86
Not completed — Lost to Follow-up | 86
Not completed — Adverse Event | 42
Not completed — Withdrawal by Subject | 41
Not completed — Other | 14
Not completed — Other | 13
Not completed — AE and Withdrew Consent | 5
Not completed — Withdrew Consent and Lack of Efficacy | 5
Not completed — Withdrew consent and Other Reason | 4
Not completed — AE and Lack of Efficacy | 4
Not completed — Death | 1
Not completed — AE and Lost to Follow-up | 1
Not completed — AE and Other Reason | 1
Not completed — AE, Withdrew Consent & Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Humira
Number analyzed (Participants) | 566
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 456
  Male | 110
Region of Enrollment [Number; unit: participants]
  Greece | 566

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
  If an adverse event meets any of the following criteria, it is considered a serious adverse event (SAE): Results in death, is life-threatening, results in hospitalization or the prolongation of hospitalization, is a congenital anomaly or a persistent or significant disability/incapacity, is an event that results in a condition that substantially interferes with the activities of daily living of the participant, is an important medical event requiring medical or surgical intervention to prevent a serious outcome, spontaneous abortion or miscarriage experienced by the participant, or an elective abortion performed on the participant.
Time Frame: 3 years
Population: The safety population, including all patients that received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 566
participants
  Any Adverse Event | 262
  Serious Adverse Event | 65

2. Primary Outcome: Disease Activity Score (DAS) 28 Over Time
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Safety population; "n" indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 566
units on a scale
  Baseline (n=555) | 6.0 (1.2)
  Month 3 (n=510) | 4.2 (1.4)
  Month 6 (n=449) | 3.8 (1.5)
  Month 9 (n=401) | 3.5 (1.5)
  Month 12 (n=379) | 3.5 (1.5)
  Month 18 (n=333) | 3.3 (1.5)
  Month 24 (n=298) | 3.2 (1.5)
  Month 30 (n=264) | 3.0 (1.4)
  Month 36 (n=254) | 2.9 (1.4)

3. Primary Outcome: European League Against Rheumatism (EULAR) Response
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS28 score. The DAS28 score ranges from 0-10, with higher scores indicating more disease activity.
  A Good EULAR Response is defined as an improvement (decrease) in the DAS28 of > 1.2 compared with Baseline and attainment of a DAS28 score of ≤ 3.2.
  A Moderate EULAR Response is defined as either:
  * an improvement (decrease) in the DAS28 of > 0.6 and ≤ 1.2 from Baseline and attainment of a DAS28 score of ≤ 5.1, or
  * an improvement (decrease) in the DAS28 of > 1.2 from Baseline and attainment of a DAS28 score of > 3.2.
  No Response is defined as either:
  * an improvement (decrease) in the DAS28 of ≤ to 0.6, or
  * an improvement (decrease) in the DAS28 of > 0.6 and ≤ 1.2 and attainment of a DAS28 of > 5.1.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Safety population;
Measure: Number; unit: participants
Groups:
- Good Response: Rheumatoid Arthritis patients treated with Humira (adalimumab) with a Good Response per EULAR criteria.
- Moderate Response: Rheumatoid Arthritis patients treated with Humira (adalimumab) with a Moderate Response per EULAR criteria.
- No Response: Rheumatoid Arthritis patients treated with Humira (adalimumab) with No Response according to EULAR criteria.
Arm/Group | Good Response | Moderate Response | No Response
Number analyzed (Participants) | 566 | 566 | 566
participants
  Month 3 (n=501) | 112 | 242 | 147
  Month 6 (n=443) | 154 | 193 | 96
  Month 9 (n=394) | 173 | 147 | 74
  Month 12 (n=373) | 171 | 139 | 63
  Month 18 (n=327) | 168 | 105 | 54
  Month 24 (n=294) | 169 | 84 | 41
  Month 30 (n=262) | 155 | 78 | 29
  Month 36 (n=253) | 156 | 68 | 29

4. Primary Outcome: Number of Participants With an American College of Rheumatology (ACR) 20 Response
Description: American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-reactive protein [CRP]).
Time Frame: Baseline and Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Safety population; the analysis was performed on the basis of non-missing information and no imputation methods were used. "n" indicates the number of patients for whom ACR20 could be calculated at each time point.
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 566
participants
  Month 3 (n=491) | 265
  Month 6 (n=427) | 279
  Month 9 (n=384) | 263
  Month 12 (n=363) | 248
  Month 18 (n=330) | 241
  Month 24 (n=293) | 216
  Month 30 (n=259) | 198
  Month 36 (n=248) | 194

5. Primary Outcome: Number of Participants With an American College of Rheumatology (ACR) 50 Response
Description: American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-reactive protein [CRP]).
Time Frame: Baseline and Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Safety population; the analysis was performed on the basis of non-missing information and no imputation methods were used. "n" indicates the number of patients for whom ACR50 could be calculated at each time point.
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 566
participants
  Month 3 (n=498) | 134
  Month 6 (n=433) | 188
  Month 9 (n=388) | 205
  Month 12 (n=368) | 182
  Month 18 (n=333) | 184
  Month 24 (n=291) | 170
  Month 30 (n=256) | 161
  Month 36 (n=250) | 164

6. Primary Outcome: Number of Participants With an American College of Rheumatology (ACR) 70 Response
Description: American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * Acute phase reactant value (C-reactive protein [CRP]).
Time Frame: Baseline and Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Safety population; the analysis was performed on the basis of non-missing information and no imputation methods were used. "n" indicates the number of patients for whom ACR70 could be calculated at each time point.
Measure: Number; unit: participants
Arm/Group | Humira
Number analyzed (Participants) | 566
participants
  Month 3 (n=495) | 67
  Month 6 (n=435) | 118
  Month 9 (n=390) | 147
  Month 12 (n=373) | 142
  Month 18 (n=330) | 154
  Month 24 (n=294) | 149
  Month 30 (n=261) | 139
  Month 36 (n=253) | 144

7. Secondary Outcome: Percentage of Participants Who Missed at Least One Dose of Humira
Description: Compliance to study treatment was measured by the percentage of participants who missed at least one dose of Humira during each time interval between study visits.
Time Frame: Months 3, 6, 9, 12, 18, 24, 30, and 36
Population: Safety population; "n" indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Humira
Number analyzed (Participants) | 566
percentage of participants
  Month 3 (n=512) | 6.6
  Month 6 (n=451) | 8.6
  Month 9 (n=406) | 7.4
  Month 12 (n=384) | 7.3
  Month 18 (n=341) | 8.2
  Month 24 (n=303) | 7.6
  Month 30 (n=271) | 5.5
  Month 36 (n=262) | 4.2

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Humira
Serious Adverse Events (participants affected / at risk) | 65/566
Other Adverse Events (participants affected / at risk) | 109/566
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=566)
Anemia (Blood and lymphatic system disorders) | 2
Lymph nodes enlarged (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Acute myocardial infarction/Myocardial infarction (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure aggravated (Cardiac disorders) | 1
Paroxysmal upraventricular tachycardia (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Abdominal bloating (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis ulcerative aggravated (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Epigastric pain (Gastrointestinal disorders) | 1
Fistula (Gastrointestinal disorders) | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 1
Hypochondrium pain right (Gastrointestinal disorders) | 1
Hypogastric pain (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatic disorder (Gastrointestinal disorders) | 1
Paresthesia circumoral (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever/Pyrexia (General disorders) | 7
Weakness/Asthenia (General disorders) | 4
Fatigue (General disorders) | 2
Difficulty in walking (General disorders) | 1
Drug ineffective (General disorders) | 1
Edema abdomen (General disorders) | 1
Edema of legs (General disorders) | 1
Nodule on finger (General disorders) | 1
Pain (General disorders) | 1
Reaction unevaluable (General disorders) | 1
Swelling (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Gallbladder perforation (Hepatobiliary disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Respiratory tract infection (Infections and infestations) | 3
Viral infection (Infections and infestations) | 2
Abscesses of skin (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Periapical dental abscess (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Phlegmon (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Post operative infection (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Relapsing fever (Infections and infestations) | 1
Septic arthritis (Infections and infestations) | 1
Tuberculous peritonitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral hepatitis B (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 5
Automobile Accident (Injury, poisoning and procedural complications) | 1
Bimalleolar fracture (Injury, poisoning and procedural complications) | 1
Elbow fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1
Shoulder fracture (Injury, poisoning and procedural complications) | 1
Weight Loss/Weight decreased (Investigations) | 2
Creatine increased (Investigations) | 1
Erythrocyte sedimentation rate increased (Investigations) | 1
Hematocrit decreased (Investigations) | 1
Transaminases increased/Hepatic enzyme increased (Investigations) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
RA flare up (Musculoskeletal and connective tissue disorders) | 4
Pain in hip (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthritis single joint (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hydrarthrosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 1
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Periarticular disorder (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Wrist deformity (Musculoskeletal and connective tissue disorders) | 1
Acute myelomonocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Collecting duct renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian germ cell cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parathyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemorrhagic stroke (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 2
Demyelinating disease (excl. multiple sclerosis) (Nervous system disorders) | 1
Movements reduced (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1
Hair loss (Skin and subcutaneous tissue disorders) | 1
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Fusion lumbar spine (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Removal of surgical hardware (Surgical and medical procedures) | 1
Abdominal aortic aneurysm (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=566)
Drug ineffective (General disorders) | 91
Respiratory infection (Infections and infestations) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.